CLINICAL TRIAL: NCT03811197
Title: Efficacy of Medical Nutrition Therapy of Obese Patients Supported by Hypnotic Suggestions or Telemedicine
Brief Title: Efficacy of Diet and Hypnotic Suggestions or Telemedicine in Obesity Management
Acronym: TASTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Warsaw University of Life Sciences (Other)
Responsible Party: Principal Investigator, Danuta Gajewska, Principal Investigator, Adjunct Professor at the Department of Dietetics,PhD, Warsaw University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hipnoza2019
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight Loss; Telemedicine; Hypnotic Suggestions
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- individual MNT (Experimental): Dietary counseling via face to face meeting
  Interventions: Behavioral: Dietary counseling via face to face meeting
- Individual MNT and T (Experimental): Dietary counseling via face to face meeting and Telemedicine
  Interventions: Behavioral: Dietary counseling via face to face meeting; Behavioral: Telemedicine
- Individual MNT and HS (Experimental): Dietary counseling via face to face meeting and Hypnotic Suggestions
  Interventions: Behavioral: Dietary counseling via face to face meeting; Behavioral: Hypnotic Suggestions

INTERVENTIONS:
Behavioral: Dietary counseling via face to face meeting — All subjects received individual MNT and individual dietary recommendations based on DASH (Dietary Approaches to Stop Hypertension) diet plan for 6 months (Part A). Dietary counseling is provided by a trained dietitian. Months 9 and 12 - follow up (Part B).
Behavioral: Telemedicine — All subjects received an additional dietary counseling for 6 months (via internet, messenger or telephone) two weeks after each standard visit will be added to the counseling (Part A). Standard and additional dietary counseling (T) are provided by a trained dietitian. Months 9 and 12 - follow up (Part B).
  Arms: Individual MNT and T
Behavioral: Hypnotic Suggestions — All subjects received individual hypnotic suggestion (HS) for 6 months as a supplementary method for dietary counseling. HS will be adapted to the "small steps" method used in the management of obesity. During the visit, HS will be recorded and the individual will listen to it every day (Part A). HS will be provided by a physician, qualified in the field of hypnotherapy. Months 9 and 12 - follow up (Part B).
  Arms: Individual MNT and HS

SUMMARY:
The aim of the study is the assessment of the effectiveness of medical nutrition therapy (MNT) among obese patients, including a well-balanced low-calories diet, an individual dietary counseling conducted by dietitians and supported by telemedicine (T) or hypnotic suggestions (HS).

The study will cover a group of 90 adult patients, both sexes, with obesity (BMI ≥30 kg/m^2) undergoing MNT a dietetic treatment. Three arms are planned in the study scheme, according to the scheme: Group 1 - individual MNT (30 people); Group 2 -individual MNT and T (30 people); Group 3 - individual MNT and HS (30 people).

The authors hope that the results of the study will allow to develop a new model of the most effective management of obesity, resulting in weight reduction and maintaining this effect over time. The results obtained during the study will also allow to assess the impact of the therapy applied on lifestyle changes, dietary habits and the knowledge about the disease among obese patients.

DETAILED DESCRIPTION:
This is a prospective randomized control trial among obese subjects. The scope of the study includes: identification of nutritional habits leading to obesity; assessment of patient's motivation to introduce life style changes; assessment of anthropometric parameters, body composition, arterial stiffness and resting metabolic rate at baseline and at specific control points; development of individual medical nutrition therapy (MNT) and weight reduction plan depending on the initial body weight of the subjects; quantitative and qualitative assessment of the diet at baseline and in each month for a period of 6 months (Part A) and 9, 12 months (Part B); assessment of nutritional knowledge at baseline and at specific control points; education of patients using the behavioral-cognitive method, conducted for 6 months; introduction of hypnotic suggestion (HS) or telemedicine (T) to support the achievement and the maintenance of the lifestyle changes.

The study covers a group of 90 adults, both sexes, with obesity (BMI ≥30 kg/m^2), undergoing individual MNT, randomly assigned to one of three groups for 6 months (Part A): Group 1 - individual MNT (30 people); Group 2 - individual MNT and T (30 people); Group 3 - individual MNT and HS (30 people). All subjects will continue the program for additional 6 months (Part B follow up).

The selection of subjects for the study is purposeful and the participation in the study is voluntary. All subjects are educated to follow a reduced calorie Dietary Approaches to Stop Hypertension diet ("DASH") for 6 months (Part A). Education materials (handouts and sample meal plans) are provided to the subjects.

The primary and secondary outcomes will be evaluated at baseline, months 1,2,3,4,5, 6 (Part A) and months 9, 12 (Part B follow up).

ELIGIBILITY:
Inclusion Criteria:

* Subject is over 18 years.
* Subject is diagnosed with obesity (BMI ≥ 30 kg / m^2 at the screening visit).
* Subject understands the study procedures and is able to give written informed consent.

Exclusion Criteria:

* Subject is under 18 years.
* Subject is a pregnant women or a breast-feeding mother; or subject is planning to be pregnant during the study period
* Subject is suffering from chronic liver diseases or renal failure
* Subject has untreated or uncompensated thyroid diseases
* Subject has a history of presence of mental disorders
* Subject has a history of presence of epilepsy
* Subject has a history of presence of cancer
* Any other uncontrolled physical or psychological condition that increases significantly the health risks for the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Body Weight | 6 months (Part A); up to 12 months (Part B)
  Changes in body weight from baseline (month 0) to each post-randomization visit (month 1, 3, 6 for Parts A and 9, 12 months for Part B)
Body Mass Index | 6 months (Part A); up to 12 months (Part B)
  Changes in BMI from baseline (month 0) to each post-randomization visit (month 1, 3, 6 for Parts A and 9, 12 months for Part B)

SECONDARY OUTCOMES:
Waist circumference | 6 months (Part A); up to 12 months (Part B)
  Changes in waist circumference from baseline (month 0) to each post-randomization visit (month 1, 3, 6 for Parts A and 9, 12 months for Part B)
Hip circumference | up to 6 months (Part A); up to 12 months (Part B)
  Changes in hip circumference from baseline (month 0) to each post-randomization visit (month 1, 3, 6 for Parts A and 9, 12 months for Part B)
Arm circumference | 6 months (Part A); up to 12 months (Part B)
  Changes in arm circumference from baseline (month 0) to each post-randomization visit (month 1, 3, 6 for Parts A and 9, 12 months for Part B)
Body composition | 6 months (Part A); up to 12 months (Part B)
  Changes in body fat mass, fat free mass, muscle mass using bioelectrical impedance analysis from baseline (month 0) to each post-randomization visit (month 1, 3, 6 for Parts A and 9, 18 months for Part B)
Health related quality of life | baseline, month 6, 9, 12
  Changes in Health related quality of life using the EQ-5D-5L questionnaire
Dietary intake | 6 months (Part A); up to 12 months (Part B)
  Changes in dietary intakes using 4-day recorded diet diaries from baseline (month 0) to each post-randomization visit
Sleep behaviour | baseline and month 6 for Parts A and month 12 for Part B
  Sleep behaviour using Athens Insomnia Scale (AIS)
Subjective assessment of health status | baseline and month 6 for Parts A and month 12 for Part B
  Changes in subjective assessment of health status using 5-points Likert-type rating scale

OTHER OUTCOMES:
Arterial stiffness | baseline, month 12
  Arterial stiffness measurement using an applanation tonometer (Sphygmocor, AtCor Medical, Sydney, Australia
Resting Metabolic Rate | baseline, month 12
  Resting Metabolic Rate measurement using FitMate metabolic system (Cosmed, Rome, Italy)
Nutritional knowledge score baseline | baseline, month 6
  Nutritional knowledge measurement using Nutritional Knowledge 13-items Test
The patient's readiness for making changes | baseline
  The patient's readiness for making changes assessed by a questionnaire (Intrinsic Motivation Inventory, IMI-SR Motivation Questionnaire) and the scale of perception of own competences

CONTACTS AND LOCATIONS:
Overall Officials: Danuta Gajewska, PhD, Principal Investigator — Department of Dietetics, Warsaw University of Life Sciences
Locations (1):
- Faculty of Human Nutrition and Consumer Sciences of the Warsaw University of Life Sciences, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided